CLINICAL TRIAL: NCT05059418
Title: Burning Mouth Syndrome - Optimized Diagnostic Criteria and Treatment
Brief Title: Burning Mouth Syndrome - New Diagnostic Criteria and Treatment
Acronym: BMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Malmö University (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Per Alstergren, Professor, Pro Dean, Malmö University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BMS001
Record Dates: First submitted 2021-08-31; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Burning Mouth Syndrome
Keywords: BMS; Chronic pain; Pain-related disability; Somatosensory changes; clonazepam; capsaicin; oral mucosa
MeSH Terms: conditions — Burning Mouth Syndrome; Chronic Pain | interventions — Clonazepam; Capsaicin

STUDY DESIGN:
Intervention Model Description: N-of-1 design. Three two-week treatment arms with a one-week wash-out period in between. After that, the patient will chose their preferred treatment and continue with that treatment for 6 months (i.e. this part is not randomized or controlled).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: One clinical examinator for all examinations (baseline examination, outcome assessments), randomization, allocation and drug management by another person,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clonazepam (Active Comparator): Topical treatment of oral mucosa with a 3-min lozenge tablet with clonazepam (0.5 mg), three times a day.
  Interventions: Drug: Clonazepam 0.5 MG
- Capsaicin (Active Comparator): Topical treatment of oral mucosa with capsaicin rinsing solution (XXXX IE) for three min three times a day.
  Interventions: Drug: Capsaicin Topical
- Placebo (Placebo Comparator): Topical treatment of oral mucosa with rinsing solution without capsaicin for three min three times a day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Clonazepam 0.5 MG — Topical treatment of oral mucosa with lozenge pill
  Other Names: Iktorivil
  Arms: Clonazepam
Drug: Capsaicin Topical — Topical treatment of oral mucosa with capsaicin rinse
  Other Names: Chili
  Arms: Capsaicin
Other: Placebo — Mouth rinse with no capsaicin
  Other Names: Inget
  Arms: Placebo

SUMMARY:
The first part of this study is to optimize diagnostic criteria for BMS, i.e. not a clinical trial, and will not be covered in this application.

The second part will compare topical treatment with clonazepam, capsaicin and placebo in a n-of-1 study design regarding effects of pain, pain-related disability, somatosensory changes in the trigeminal nerve and patient experience in patients with primary BMS or other oral mucosal pain. The patients will be treated for two weeks with each drug, with a one-week wash-out period in between. After the last washed-out period, the patients will be able to chose the treatment that they prefer the most and continue with that treatment during 6 months.

DETAILED DESCRIPTION:
The clinical trial in the present study will investigate treatment effects on pain, pain-related disability, jaw function and patients' experiences by topical treatment with clonazepam or capsaicin in comparison with placebo in patients with BMS or other oral mucosal pain.

Twenty patients with primary BMS and 20 patients with other oral mucosal pain will be included. The study will comprise a n-of-1-design where each participant will be it's own control.

The study will compare topical treatment with clonazepam, capsaicin and placebo regarding effects of pain, pain-related disability, somatosensory changes in the trigeminal nerve and patient experience. primary outcome will be pain intensity and patient experience.

The patients will be treated for two weeks with each drug, with a one-week wash-out period in between. After the last washed-out period, the patients will be able to chose the treatment that they prefer the most and continue with that treatment during 6 months. After this 6 months, pain, pain-related disability, somatosensory changes in the trigeminal nerve and patient experience will be assessed again.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary BMS according to International Classification of Orofacial Pain (ICOP) OR diagnosis of other oral mucosal pains according to ICOP

Exclusion Criteria:

* Fibromyalgia
* IBS
* Reflux
* Recent (<3 months) intraoral surgical procedure
* Ongoing medication with Clonazepam or Capsaicin

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Point measurement, will be assessed immediately before start of treatment
  Overall oral mucosa pain intensity. Will be assessed using the subscale "Characteristic pain intensity" (three numerical rating scales 0 - 10 assessing current pain. intensity as well as worst and average pain intensity during the last two weeks) in the Graded Chronic Pain Scale
Pain intensity | Point measurement, will be assessed 10 days after treatment start for each treatment period.
  Overall oral mucosa pain intensity. Will be assessed using the subscale "Characteristic pain intensity" (three numerical rating scales 0 - 10 assessing current pain. intensity as well as worst and average pain intensity during the last two weeks) in the Graded Chronic Pain Scale
Pain intensity | Point measurement, will be assessed the day after each treatment period is finished (22 days after start of each treatment)
  Overall oral mucosa pain intensity. Will be assessed using the subscale "Characteristic pain intensity" (three numerical rating scales 0 - 10 assessing current pain. intensity as well as worst and average pain intensity during the last two weeks) in the Graded Chronic Pain Scale
Patient satisfaction | Point measurement, will be assessed immediately before start of treatment
  Patient satisfaction with the treatment tested. Will be assessed using a numerical rating scale 0 - 10 where 0 = very dissatisfied and 10 = very satisfied.
Patient satisfaction | Point measurement, will be assessed 10 days after treatment start for each treatment period.
  Patient satisfaction with the treatment tested. Will be assessed using a numerical rating scale 0 - 10 where 0 = very dissatisfied and 10 = very satisfied.
Patient satisfaction | Point measurement, will be assessed the day after each treatment period is finished (22 days after start of each treatment)
  Patient satisfaction with the treatment tested. Will be assessed using a numerical rating scale 0 - 10 where 0 = very dissatisfied and 10 = very satisfied.

SECONDARY OUTCOMES:
Pain-related disability | Point measurement, will be assessed immediately before start of treatment as well as one, two and three weeks after treatment start.
  Pain-related disability from oral mucosal pains. Will be assessed using the subscale "Pain-related Disability" (three numerical rating scales 0 - 10 assessing impact on the oral pain on general, social and work-related activities during the last two weeks) in the Graded Chronic Pain Scale

CONTACTS AND LOCATIONS:
Overall Officials: Per Alstergren, PhD, Prof, Principal Investigator — Malmö University

IPD SHARING:
Plan to Share IPD: No